CLINICAL TRIAL: NCT06342219
Title: Study Protocol for a Randomized Controlled Trial of Neurofeedback Mindfulness in Chronic Migraines
Brief Title: Chronic Migraines and Neurofdeeback Mindfulness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (Other)
Responsible Party: Principal Investigator, Marla Mickleborough, Dr. Marla Mickleborough, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 423629
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Chronic Migraine, Headache
Keywords: neurofeedback mindfulness; headache management self-efficacy; chronic migraines; dependence behaviours; migraine severity
MeSH Terms: conditions — Headache

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- neurofeedback mindfulness (Experimental): This group is asked to do 10 min/day practice of neurofeedback mindfulness for 8 weeks. They should sit comfortably in a quiet area and do one of ten beginner self-guided mindfulness sessions on mind-body scanning techniques from within the MUSE app. Each session includes a brief explanation for 2-3 minutes before the practice. Once the participants start their practices, they receive sounds for their real-time brain activities: thunderstorm for an active state, ocean waves for a neutral state, and birds chirping for a relaxed state. For each five seconds of consistent relaxed state, the participants are reinforced with points.
  Interventions: Behavioral: Neurofeedback Mindfulness
- Attention Task (Active Comparator): The participants in the controlled intervention group are assigned to have an attention routine in a relaxed position. They are required to sit comfortably and relax in a quiet area to put on their MUSE headband, set it up, and use the same practices on MUSE app but they will mute all the neurofeedback sounds and instructions. Instead, on their smartphone the participants will check their emails, the news, or their preferred social media platform for 10 minutes. Once the session is over, the participants receive the graphical feedback of their brain activities. The feedback includes a timeline indicating their brain states (active, or relaxed) during the 10-minute session.
  Interventions: Behavioral: Attention Task
- Waitlisted Group (No Intervention): The participants in this group are informed about being appointed in the waitlisted group and that we will only be collecting headache data from them for 8 weeks. They will complete the questionnaires for three rounds (i.e., Week 1, Week 4, and Week 8) and information about their headaches will be collected via the headache diaries. After 8 weeks, they will receive the MUSE device and will be offered a complementary session on how to use the device for their personal use. A debriefing form will be emailed to all the participants after completion of the study.

INTERVENTIONS:
Behavioral: Neurofeedback Mindfulness — The participants will use a portable EEG headband (MUSE) which is a noninvasive tool for collecting EEG data. They will receive real-time EEG data given an audio feedback while doing their daily mindfulness practice.
  Arms: neurofeedback mindfulness
Behavioral: Attention Task — The participants in this arm will use the portable EEG while listening to an audiobook. They will receive a summary of their brain activities after task completion on each day.
  Arms: Attention Task

SUMMARY:
As the second phase of our study on migraine headaches and neurofeedback mindfulness, we will explore how chronic migraineurs will benefit from a long term practice (8 weeks) of neurofeedback mindfulness compared to a similar attention group and a waitlisted group. This randomized controlled trial will also explore if migrianuers could decrease their dependence on medicine intake after completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of chronic migraine from a clinician or have met the criteria for a chronic migraine diagnosis based on ICHD-3
* reside in Saskatoon area
* have a smartphone and internet connection for accessing the MUSE app
* have no frequent background experience of meditation

Exclusion Criteria:

* Comorbidity of Raynaud's syndrome or diabetes
* Current use of a preventative migraine treatment over 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Migraine Disability | 8 weeks
  measured by Migraine Disability Assessment Scale (MIDAS)
Migraine Severity | 8 weeks
  measured by Headache Impact Test-short form (HIT-6)
Headache management self-efficacy | 8 weeks
  measured by Headache Management Self-Efficacy Scale
Dependence on medicine | 8 weeks
  measured by Severity of Dependence Scale (SDS)

SECONDARY OUTCOMES:
Anxiety | 8 weeks
  measured by BECK Anxiety Inventory (BAI)
Depression | 8 weeks
  measured by The Center for Epidemiologic Studies Depression (CES-D)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No